CLINICAL TRIAL: NCT07118163
Title: The Relationship Pain Beliefs With Kinesiophobia, Catastrophizing, Pain Knowledge, and Disability in Individuals With Shoulder Pain
Brief Title: The Relationship Pain Beliefs With Kinesiophobia, Catastrophizing, Pain Knowledge, and Shoulder Functional Disability in Individuals With Shoulder Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, MSc. PT., Istanbul University - Cerrahpasa
Other Study IDs: IUC25
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain Chronic; Impingement Syndrome
Keywords: Rotator cuff; Shoulder Pain; Organic Pain Beliefs
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with shoulder pain
  Interventions: Other: Other; Other: No intervention; Observational study

INTERVENTIONS:
Other: Other — No intervention was applied in this study.
Other: No intervention; Observational study — No intervention

SUMMARY:
This cross-sectional observational study aims to examine the relationship between psychological and organic pain beliefs and kinesiophobia, pain catastrophizing, pain knowledge, and shoulder functional disability (SPADI) in individuals with shoulder pain. The study seeks to clarify how pain-related beliefs influence physical and psychological outcomes in musculoskeletal shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 75 years
* Presence of shoulder pain for at least 3 months
* At least one positive finding in each of the following categories:
* Painful arc during flexion or abduction
* Positive Neer's or Kennedy-Hawkins tests
* Pain during resisted external rotation, abduction, or empty can test

Exclusion Criteria:

* History of shoulder dislocation or fracture in the past 12 months
* Presence of full-thickness rotator cuff tear
* Previous shoulder surgery
* Received physiotherapy or corticosteroid injection for the shoulder in the past 3 months
* Presence of adhesive capsulitis (passive shoulder range of motion < 50%)
* Presence of systemic diseases such as cancer or rheumatic disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes individuals aged between 18 and 75 who present with shoulder pain and seek care at a healthcare facility. Participants must have sufficient cognitive ability to complete the questionnaires independently. Participation in the study will be on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain Beliefs | Baseline
  To examine how psychological and organic pain beliefs

SECONDARY OUTCOMES:
Kinesiophobia | Baseline
  To examine fear of movement
Catastrophizing | Baseline
  To examine tendency to catastrophize pain experiences.
Pain Knowledge | Baseline
  To examine level of knowledge and understanding of pain neurophysiology
Shoulder Pain and Disability Index (SPADI) | Baseline
  To examine the disability level of patients

IPD SHARING:
Plan to Share IPD: Undecided